CLINICAL TRIAL: NCT05103475
Title: Rage Against the Pain: An Alternative Yoga Program to Address Chronic Low Back Pain Among Veterans
Brief Title: Rage Against the Pain to Address Chronic Low Back Pain Among Veterans
Acronym: RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 19-362
Record Dates: First submitted 2021-10-01; First posted 2021-11-02 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Yoga; Veterans; Complementary and integrative health
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to the RAP or control (Hatha yoga) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rage Against the Pain (RAP) (Experimental): The sets of body positions used in the RAP program will mirror those used in the Hatha Yoga classes, but the RAP program will differ from this traditional yoga practice in a number of ways: (1) the classes will be set to rock/heavy metal music; (2) meditation will not be incorporated; (3) yoga terms will not be used to describe the body positions (rather, positions will be cued in plain descriptive English terms); (4) the culminating activity for the class will be called a 'cool down' (rather than the savasana exercise typically used in yoga practice).
  Interventions: Behavioral: Rage Against the Pain (RAP)
- Control (Active Comparator): The control group will comprise a program akin to Hatha yoga with chair modifications available to all Veterans who choose/need to use them.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Rage Against the Pain (RAP) — The sets of body positions used in the RAP program will mirror those used in the Hatha Yoga classes, but the RAP program will differ from this traditional yoga practice in a number of ways: (1) the classes will be set to rock/heavy metal music; (2) meditation will not be incorporated; (3) yoga terms will not be used to describe the body positions (rather, positions will be cued in plain descriptive English terms); (4) the culminating activity for the class will be called a 'cool down' (rather than the savasana exercise typically used in yoga practice).
  Arms: Rage Against the Pain (RAP)
Behavioral: Control — The control group will comprise a program akin to Hatha yoga with chair modifications available to all Veterans who choose/need to use them.
  Other Names: Yoga
  Arms: Control

SUMMARY:
Chronic low back pain is a leading cause of disability among Veterans. Yoga is recommended as a front-line treatment option for chronic low back pain and is available across the VA healthcare system; however, despite yoga being the most widely adopted of VHA's Complementary and Integrative Health (CIH) therapies, Veteran participation in yoga still remains limited. Although it can be effective in managing pain, individuals cannot reap the benefits of yoga if they are unwilling to adopt it. One potential barrier to adoption of yoga among Veterans may be their perceptions of yoga, which for some, encompass long-held but perhaps inaccurate beliefs of what the practice entails and how their participation will be viewed by others. The goal of this study was to develop and evaluate an alternative-to-yoga program intended to improve Veteran participation and by extension, outcomes among Veterans with chronic low back pain. Based on Veteran input, we called this yoga program Rage Against the Pain (RAP) 'High Intensity Stretching'.

DETAILED DESCRIPTION:
Background: Chronic low back pain is a leading cause of disability among Veterans. Yoga is recommended as a front-line treatment option for chronic low back pain and is available across the Veterans Health Administration (VHA) healthcare system; however, despite yoga being the most widely adopted of VHA's Complementary and Integrative Health (CIH) therapies, Veteran participation in yoga still remains limited. Although it can be effective in managing pain, individuals cannot reap the benefits of yoga if they are unwilling to adopt it. One potential barrier to adoption of yoga among Veterans may be their perceptions of yoga, which for some, encompass long-held but perhaps inaccurate beliefs of what the practice entails and how their participation will be viewed by others. The goal of this study was to to develop and evaluate an alternative-to-yoga program intended to improve Veteran participation and by extension, outcomes among Veterans with chronic low back pain. Based on Veteran input, we called this yoga program Rage Against the Pain (RAP) 'High Intensity Stretching'.

Significance/Impact: The RAP program is an innovative approach to address a top priority of the VHA - using CIH therapies for pain management. The long-term goal of this work is to develop a scalable and sustainable alternative-to-yoga program for Veterans with chronic pain.

Innovation: The RAP program comprises an expressive, active practice set to music commonly enjoyed among many Veterans (e.g., rock, metal). The development of RAP (and the program name) reflects direct Veteran feedback.

Specific Aims: The Specific Aims of this project were to: (1) Develop the RAP program, which encompassed finalizing the program curriculum, including music play-lists, cues for self-expression, and sets of body positions that may be beneficial for low back pain; (2) Examine the feasibility and acceptability of offering RAP for Veterans with chronic low back pain, and; (3) Gather preliminary data to provide the foundation for process, sample size and power considerations for a future clinical trial to examine the effectiveness of RAP on Veterans' outcomes and medication use.

Methodology: We first developed the RAP program, including a home practice manual, sets of body positions, music playlists, and scripts to translate Sanskrit cuing to plain language. We then conducted a single-site pilot randomized controlled trial with two cohorts of 18 Veterans each (n=36). We randomized Veterans to the intervention (RAP) or control (Hatha yoga) group. Each cohort spanned 12 weekly one-hour sessions. We collected baseline (n=36) and follow-up (n=26) survey data and completed semi-structured interviews with a subset of survey respondents (n=20). Survey data were analyzed using bivariate comparisons. Interview transcripts were independently coded by two qualitative experts and analyzed using thematic coding techniques.

Implementation/Next Steps: We intend to conduct a larger multi-site trial of the RAP program to examine its effectiveness and issues associated with its implementation.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be eligible to participate in the study if they:

* currently receive primary care services at the Hines VA
* received a diagnosis associated with chronic low back pain in the previous 3 months

Exclusion Criteria:

Veterans will be ineligible to participate in the study if any of the following are true for them:

* they currently regularly participate in yoga
* they regularly participated in yoga in the previous 6 months
* their back pain is a symptom of a specific treatable or underlying disease/condition(s), e.g.,

  * ankylosing spondylitis
  * active or recent malignancy
  * fracture/spinal cord injury
  * spinal infection)
* they are experiencing progressive neurological deficits
* they have any other condition which results in severe disability, e.g.,

  * non-ambulatory
  * hemiparesis
  * severe cognitive deficits
* they have a diagnosis associated with psychosis
* they are currently experiencing issues around substance abuse (not including prescription opioids), as identified through ICD-10 codes associated with 'mental and behavioral disorders due to psychoactive substance use' recorded in the patient's medical record in the previous 3 months
* they do not plan to be living in the Chicagoland area for the duration of the study
* they are pregnant at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bella Etingen, PhD MA BS, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (i.e., Yoga): The control group will comprise a program akin to Hatha yoga with chair modifications available to all Veterans who choose/need to use them.
Period: Overall Study
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Started | 18 | 18
Completed (Because of the way that our primary outcomes are defined, all Veterans were included in primary outcome analyses. The definition we used for 'Completed' is the number of Veterans who completed a post-participation survey; please note that post-participation surveys were sent to all 36 Veterans who were randomized, including those who dropped out of yoga classes.) | 11 | 15
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participant age at first intervention session.
  Years | 57.0 (13.5) | 67.1 (13.8) | 62.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — As documented in the VA Corporate Data Warehouse administrative data.
  Participants
    Female | 2 | 3 | 5
    Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — As documented in the VA Corporate Data Warehouse administrative data.
  Participants
    Hispanic or Latino | 7 | 2 | 9
    Not Hispanic or Latino | 11 | 16 | 27
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — As documented in the VA Corporate Data Warehouse administrative data. Please note that we included 'Other' race with 'Unknown or Not Reported'.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 3 | 11
    White | 9 | 14 | 23
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Program Initiation (e.g., Reach)
Description: Program initiation (e.g., reach) will be defined as the number of individuals who start the RAP or Hatha yoga programs after being screened, deemed eligible for participation, and randomized to one or the other.
Time Frame: Baseline (following randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 18 | 18
Participants | 16 | 15
Statistical Analysis 1: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 1.0, Fisher Exact — The investigators used Fisher's exact due to small cell sizes; The reported value represents the calculated p-value for the Fisher's Exact test

2. Primary Outcome: Program Participation (e.g., Sustained Engagement) - Average Number of Classes Attended
Description: Program participation (e.g., sustained engagement) - average number of classes attended; this will be defined as the average number of classes Veterans attended for each respective program.
Time Frame: Post-intervention follow-up (within approximately 1 week of when the 12-week yoga or RAP programs are finished)
Measure: Mean (Standard Deviation); unit: Average number of classes attended
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 18 | 18
Average number of classes attended | 5.9 (4.9) | 4.5 (3.8)
Statistical Analysis 1: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.35, t-test, 2 sided

3. Primary Outcome: Program Participation (e.g., Sustained Engagement) - Number of Veterans Who Attend Majority of Classes
Description: Program participation (e.g., sustained engagement) - number of Veterans who attend majority of classes; this will be defined as the number of Veterans who attended the majority (9/12) of classes.
Time Frame: Post-intervention follow-up (within approximately 1 week of when the 12-week yoga or RAP programs are finished)
Measure: Count of Participants; unit: Participants
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 18 | 18
Participants | 8 | 3
Statistical Analysis 1: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.15, Fisher Exact — The investigators used Fisher's Exact due to small cell sizes

4. Secondary Outcome: Pain Intensity
Description: Pain intensity will be measured using the Defense and Veterans Pain Rating Scale, a valid and reliable numeric rating scale that asks individuals to report the average intensity of their low back pain on a scale of 0 (no pain) to 10 (worst pain imaginable) for the previous 7 days.
Time Frame: Baseline and post-intervention follow-up (within approximately 1 week of when the 12-week yoga or RAP programs are finished)
Population: Please note that, for the control group, we had baseline data for 15 individuals and follow-up data for 11 individuals.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
score on a scale
  Baseline | 5.1 (1.8) | 6.5 (1.6)
  Follow-Up: number analyzed (Participants) | 11 | 11
  Follow-Up | 4.0 (2.4) | 5.9 (1.9)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison for control group scores; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.43, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison for RAP group score; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.24, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.53, ANOVA — F = 0.41

5. Secondary Outcome: Pain Interference
Description: Pain interference (how much the individual's pain has interfered with all aspects of their life in the prior 7 days) will be measured using the validated, reliable Patient-Reported Outcomes Measurement Information System (PROMIS) 8-item pain interference short form. PROMIS scores are standardized to reflect the general adult US population, such that a mean score of 50 reflects the population mean (with a standard deviation of 10), and higher scores indicate greater levels of pain interference.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
t-score
  Baseline | 63.0 (6.3) | 64.6 (4.4)
  Follow-Up | 59.2 (6.3) | 63.8 (6.2)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison for control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.70, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison for RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.17, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.18, ANOVA — F = 1.95

6. Secondary Outcome: Back Pain-related Function
Description: Back pain-related function will be measured using the Roland-Morris Disability Questionnaire (RMDQ), a valid and reliable scale of physical disability resulting from chronic low back pain. The RMDQ asks individuals to read 24 items noting back pain-related functional impairments and mark those that describe them. All marked items are summed for a total score ranging from 0 (no impairment) to 24 (maximum impairment).
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
score on a scale
  Baseline | 10.1 (6.4) | 14.1 (5.3)
  Follow-Up | 8.5 (4.5) | 12.2 (5.9)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison - control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.37, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison - RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.50, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.90, ANOVA — F = 0.01

7. Secondary Outcome: Sleep
Description: Sleep will be measured using the Insomnia Severity Index, which is a valid and reliable 7-item scale that produces a composite score of an individual's level of sleep disturbance during the past 14 days. Item responses are added to obtain a total scale score (range: 0-28); greater scores indicate more disturbed sleep and cut-points are provided by the scale developers that map to levels of clinical severity of sleep disturbance.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
score on a scale
  Baseline | 14.5 (7.7) | 15.9 (6.8)
  Follow-up | 11.1 (8.3) | 14.5 (6.2)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison - control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.56, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison - RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.32, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.41, ANOVA — F = 0.71

8. Secondary Outcome: Depression
Description: Depression severity will be measured using the 8-item Patient Health Questionnaire (PHQ-8), a valid and reliable measure that assesses individual's depression severity by asking them to evaluate 8 items that reflect symptoms of depression and indicate how often they have experienced each in the prior two weeks on a scale of 0 to 3 (not at all - nearly every day). Scores range from 0 (no depression symptomology) to 24 (most severe symptomology); scores can also be classified into mild, moderate, moderately severe and severe categories using cut-scores defined by the scale developers.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
score on a scale
  Baseline | 9.1 (6.9) | 9.6 (4.7)
  Follow-Up | 7.6 (6.0) | 8.2 (6.4)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison - control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.50, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison - RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.60, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.98, ANOVA — F = 0.0

9. Secondary Outcome: Stress
Description: Stress will be measured using the Perceived Stress Scale (PSS) - 4 Item, a valid and reliable measure of individual's perceptions of how stressful their life experiences are. The PSS is comprised of 4 questions and produces a composite score of perceived stress (range: 0-16; higher scores indicate higher perceptions of stress).
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
score on a scale
  Baseline | 8.2 (2.9) | 7.4 (2.1)
  Follow-Up | 6.4 (2.8) | 7.9 (2.6)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison - control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.54, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison - RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.15, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.04, ANOVA — F = 4.9

10. Secondary Outcome: Use of Other Pain Management Strategies
Description: The investigators will ask participants to self-report use of other pain management activities.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Mean pain management activities reported
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
Mean pain management activities reported
  Baseline | 1.6 (1.4) | 1.7 (1.6)
  Follow-up | 2.5 (1.0) | 2.9 (2.1)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison - control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.11, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison - RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.09, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.75, ANOVA — F = 0.10

11. Secondary Outcome: Perceptions of the Program
Description: The investigators will ask participants about their perceptions of the program (extent to which they liked it, would participate again, would recommend to a peer, felt it impacted their health and how).
Time Frame: Post-intervention follow-up (within approximately 1 week of when the 12-week yoga or RAP programs are finished)
Population: These data are self-report and were gathered via separate survey questions; as such, n's may differ between questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 14
Participants
  Liked the program - extremely or quite a bit: number analyzed (Participants) | 10 | 13
  Liked the program - extremely or quite a bit | 9 | 6
  Likelihood of participating in a program like it in the future - extremely or quite a bit | 8 | 7
  Helped manage back pain - extremely or quite a bit: number analyzed (Participants) | 10 | 13
  Helped manage back pain - extremely or quite a bit | 8 | 2
  Would recommend the program to another Veteran: number analyzed (Participants) | 10 | 12
  Would recommend the program to another Veteran | 8 | 9
Statistical Analysis 1: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Likelihood to participate in a program like it in the future; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.41, Fisher Exact; The investigators used Fisher's Exact due to small cell sizes
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Help to manage back pain; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.003, Fisher Exact — The investigators used Fisher's Exact due to small cell sizes
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Would recommend to another Veteran; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 1.00, Fisher Exact — The investigators used Fisher's Exact due to small sample sizes; The reported value represents the calculated p-value for the Fisher's Exact test
Statistical Analysis 4: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); Liked the program; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.07, Fisher Exact — The investigators used Fisher's Exact due to small cell sizes

12. Secondary Outcome: Pain Medication Use
Description: The investigators will ask participants to self-report any pain medication use.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Average number of medications reported
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
Number analyzed (Participants) | 11 | 15
Average number of medications reported
  Baseline | 2.3 (2.1) | 2.5 (1.8)
  Follow-Up | 1.7 (1.7) | 2.4 (1.4)
Statistical Analysis 1: Comparison: Control (i.e., Yoga); Pre/post comparison - control group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.91, t-test, 2 sided
Statistical Analysis 2: Comparison: Rage Against the Pain (RAP); Pre/post comparison - RAP group; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.51, t-test, 2 sided
Statistical Analysis 3: Comparison: Rage Against the Pain (RAP) vs Control (i.e., Yoga); ANOVA results - group x time interaction; Test type: Other — Please note that all data analyses were exploratory because this was feasibility pilot; p = 0.42, ANOVA — F = 0.68

ADVERSE EVENTS:
Time Frame: 24 weeks total (12 weeks per group for each cohort).
Arm/Group | Rage Against the Pain (RAP) | Control (i.e., Yoga)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05103475/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT05103475/ICF_002.pdf